CLINICAL TRIAL: NCT03679507
Title: The Effect of Low Intensity Ultrasound Therapy on Chronic Pain Due to Osteoarthritis of the Knee.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dr. Kevin Rod (Other)
Responsible Party: Sponsor-Investigator, Dr. Kevin Rod, Director, Toronto Poly Clinic
Organization: Toronto Poly Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TPC-5460-204-0918
Record Dates: First submitted 2018-09-13; First posted 2018-09-20 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Osteoarthritis in the Knee

STUDY DESIGN:
Intervention Model Description: This clinical trial will investigate the safety and efficacy of a new hand-held, low-intensity therapeutic ultrasound (LIPUS) device to treat chronic knee pain in osteoarthritis patients. Osteoarthritis of the knee is painful condition, and a leading cause of disability [11]. Two meta-analyses of this application indicate its efficacy in controlling pain [7,10]; one in improving function [10]. Three randomized, double blind, placebo-controlled studies have been published recently. Two demonstrate the ameliorative effects of low-intensity ultrasound therapy on pain, function and quality of life in patients with knee osteoarthritis [12,13]; one showed no significant difference from placebo [9]. Significantly, no adverse event was reported in any of these clinical trials. However subjects will have 24 hours phone access and email access to study administrator and study investigator for reporting any type of adverse event and seeking guidance if needed.
Who Masked: Participant, Care Provider, Investigator
Masking Description: A Study Administrator will assign subjects to a treatment group randomly, and keep this information strictly confidential. Subjects and investigators will be blinded. The Study Administrator will assign each participant a randomly generated Patient ID number to be used in the collection of data.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Active Comparator): The first patient group will receive Low Intensity Ultrasound Therapy on the affected knee joint, using the CPI-LIPUS Device
  Interventions: Procedure: Low Intensity Ultrasound Therapy
- Group B (Placebo Comparator): Will be "treated" with an identical device whose ultrasound emitting capabilities has been nullified. This device appears to operate, including illumination of the operating light.
  Interventions: Procedure: Low Intensity Ultrasound Therapy
- Group B1 (Active Comparator): The first patient group will receive high CBD oil applied topically to the affected knee joint.
  Interventions: Other: Enhancing CBD oil penetration into joints by sonophresis
- Group B2 (No Intervention): This group of patients will not receive high CBD oil to the affected joint.

INTERVENTIONS:
Procedure: Low Intensity Ultrasound Therapy — Subjects suffering from chronic pain due to osteoarthritis of the knee will be recruited for this study, and randomly assigned to two groups. One-half of these Subjects (Group A) will receive ultrasound therapy as detailed below on the affected joint; the other half (Group B) is a placebo group.
  Arms: Group A; Group B
Other: Enhancing CBD oil penetration into joints by sonophresis — High CBD oil will be applied to the affected knee of one-half of the recruited subjects.
  Arms: Group B1

SUMMARY:
To evaluate a new, low intensity ultrasound device in the treatment of chronic pain due to osteoarthritis in the knee.

Enhancing CBD oil penetration into joints by sonophoresis.

DETAILED DESCRIPTION:
Materials and Methods:

Inclusion criteria:

1. Osteo-arthritis of knee joint diagnosed through X-Ray evaluation
2. Moderate or sever level of pain due to knee osteoarthritis and no other known reason
3. Male of Female patients of 18 to 85 years old
4. Pain interfering with activities of daily life

Exclusion criteria:

1. Cancer pain or any other concurrent cancerous condition
2. History of Knee replacement surgery in the study joint
3. Local infection or any kind of inflammatory or allergic skin lesion
4. Rheumatoid arthritis
5. Mobility disorders or not being able to walk

Subjects suffering from chronic pain due to osteoarthritis of the knee will be recruited for this study, and randomly assigned to two groups. One-half of these Subjects (Group A) will receive ultrasound therapy as detailed below on the affected joint; the other half (Group B) is a placebo group. Assuming 60% of subjects in Group A show some improvement, as do 30% of patients in Group B, total enrolment of 84 patients (42 per group) will yield statistically significant results (p=0.05; 80% power).

A Study Administrator will assign subjects to a treatment group randomly, and keep this information strictly confidential. Subjects and investigators will be blinded. The Study Administrator will assign each participant a randomly generated Patient ID number to be used in the collection of data.

Subjects will provide in advance written consent to participate in the study, in accordance with Health Canada requirements. Participating subjects will provide baseline pain assessments prior to their first treatment using a 10-point Numeric Pain Scale. They will indicate their current level of pain, and the best and worst pain experienced in the previous 24 hours. An average of these three ratings will be noted. Additionally, participants will complete a Brief Pain Inventory, indicating the location(s) of their pain as well as its impact on general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life.

Group A: The first patient group will receive ultrasound therapy on the affected knee joint, using the CPI-LIPUS Device (Circuit Plus Inc., Richmond Hill, Ontario). This low intensity pulsed ultrasonic system operates at 1 MHz for a fixed time of 5 minutes, with a pulsed repetition of 1 kHz. Its total acoustic power is 6.3 W 5%, equivalent to 1.2 W/cm2 acoustic intensity. (Complete technical specifications of and instructions for CPI-LIPUS are attached as Appendix I.) Ultrasound treatment will be pulsed at 50%.

The head of device will be applied to the most painful area of the knee (typically the medial or lateral upper quadrant) for one cycle of five minutes using ultrasound conductive media providing rotating movements, applying only enough pressure to provide adequate coupling of treatment head and the treatment area.

Group B: Group B will be "treated" with an identical device whose ultrasound emitting capabilities has been nullified. This device appears to operate, including illumination of the operating light. The head of the device will be applied to the most painful area of the knee (typically the medial or lateral upper quadrant) for five minutes exactly in the same manner as the Group A.

Treatment of all patients will take place at Toronto Poly Clinic, Toronto Ontario, a multi-disciplinary clinic focused on the treatment of chronic pain. Lead investigator Dr. Rod is their treating physician. Treatments will be repeated at an interval of seven days. A total of six treatments will be performed. Pain assessments will be conducted prior to each treatment, and at 14 days following the last treatment.

Toronto Poly Clinic follows the College of Physicians and Surgeons of Ontario practice regulations including confidentiality and privacy rules and regulations. Study materials will only have subject/patient ID number.

Participating patients will have free access to their usual analgesic treatments throughout the study. A condition of participation in the trial is the patients' agreement to maintain their current analgesic regimen, without change in medication or dosage.

Once a day, participating subjects will rate their joint pain and ease of use of the joint on 10-point Likert scales. They will also record any use of analgesic medication. These data will be noted in Patient Diaries, whose only identifier will be the Patient ID number for maintaining full confidentiality and privacy.

Data from pain assessments, and from the Patient Diaries, will be analyzed to determine the impact of ultrasound therapy on chronic pain due to osteoarthritis of the knee joint. Statistical significance will be assessed.

Data safety: All study materials, diaries, assessments and clinical notes collectively called data will be kept in secure server of the clinic for electronic data or locked cabinet of a secure area in clinic for paper data documents.

ELIGIBILITY:
Inclusion Criteria:

1. Osteo-arthritis of knee joint diagnosed through X-Ray evaluation
2. Moderate or sever level of pain due to knee osteoarthritis and no other known reason
3. Male of Female patients of 18 to 85 years old
4. Pain interfering with activities of daily life

Exclusion Criteria:

1. Cancer pain or any other concurrent cancerous condition
2. History of Knee replacement surgery in the study joint
3. Local infection or any kind of inflammatory or allergic skin lesion
4. Rheumatoid arthritis
5. Mobility disorders or not being able to walk

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Measure | The outcome will be measured over a period of 6 weeks.
  Participants who receive treatment using the CPI-LIPUS , a low intensity pulsed ultrasonic device will document any changes to their pain severity on a Brief Pain Inventory numeric scale from 1 to 10, with 1 being no pain, and 10 being the worst pain at each appointment.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Poly Clinic, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No